CLINICAL TRIAL: NCT01104168
Title: Diabetes Care in Nursing Home Residents
Brief Title: Diabetes in the Elderly: Retrospective Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Other Study IDs: IRB00035147
Record Dates: First submitted 2010-04-09; First posted 2010-04-15 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes
Keywords: diabetes; elderly; nursing home resident
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nursing home residents with diabetes

SUMMARY:
Diabetes is highly prevalent in the elderly, afflicting about 20% of older adults aged 65-75 years and 40% of adults >80years of age. Management of hyperglycemia is challenging in the geriatric population in long-term facilities. Numerous factors place hospitalized patients at increased risk for hyperglycemia including aging, sedentary life, stress of medical and surgical comorbidities, and changes in antidiabetic regimen. In addition, elderly patients often experience changes in their nutritional intake and organ dysfunction which increase the risk of hypoglycemic events.

There are only a few retrospective studies in elderly patients analyzing quality of diabetes care and glycemic control adjusted for medications and presence of co-morbidities in long-term care facilities. In addition, no randomized controlled trials have demonstrated benefits of glycemic control on clinical outcome, quality of life, and rate of acute metabolic complications (hyperglycemia and hypoglycemic events) in long-term care facilities.

DETAILED DESCRIPTION:
The investigators will conduct a retrospective study to determine the prevalence of diabetes, comprehensively describe the management of diabetes, and to evaluate the impact of quality of care and glycemic control on clinical outcome in elderly subjects admitted to two large long-term care facilities: Grady Health System (GHS) and Veterans Administration Medical Center (VAMC) in Atlanta, Georgia between 1/01/08 to 12/31/08.

ELIGIBILITY:
Inclusion Criteria:

* ages 65+
* diagnosis of diabetes

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older adults ages 65+ admitted to two large long-term care facilities
Sampling Method: Non-Probability Sample
Enrollment: 1409 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
prevalence of diabetes | 1 year

SECONDARY OUTCOMES:
differences in glycemic control | 1 year
  determine differences in glycemic control as measured by mean daily blood glucose concentration between different insulin regimens
evaluate the impact of quality of care and glycemic control on clinical outcome in elderly subjects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - A.G. Rhodes Homes, Atlanta, Georgia
  - Bud Terrace Homes, Atlanta, Georgia